CLINICAL TRIAL: NCT04584515
Title: A Phase I, Open-label, Fixed-Sequence Study to Evaluate the Effect of Multiple-dose Itraconazole or Rifampicin Capsules on the Single-dose PK (Pharmacokinetics) Profiles of IMP4297 Capsules in Healthy Subjects
Brief Title: IMP4297 DDI (Drug-Drug Interaction)Trial in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IMP4297-104
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — senaparib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMP4297 40 mg (Experimental): Sequential treatments of IMP4297 alone, followed by Itraconazole + IMP4297, with a washout period in between.
  Interventions: Drug: IMP4297 40 mg
- IMP4297 100 mg (Experimental): Sequential treatments of IMP4297 alone, followed by Rifampin + IMP4297, with a washout period in between.
  Interventions: Drug: IMP4297 100 mg

INTERVENTIONS:
Drug: IMP4297 40 mg — IMP4297 40 mg: IMP4297 alone, Itraconazole + IMP4297
  Other Names: Itraconazole
  Arms: IMP4297 40 mg
Drug: IMP4297 100 mg — IMP4297 100 mg: IMP4297 alone, Rifampin + IMP4297
  Other Names: Rifampin
  Arms: IMP4297 100 mg

SUMMARY:
A Phase I, Open-label, Fixed-Sequence Study to Evaluate the Effect of Multiple-dose Itraconazole or Rifampicin Capsules on the Single-dose PK Profiles of IMP4297 Capsules in Healthy Subjects

DETAILED DESCRIPTION:
Study design A Phase I, single-center, open-label, fixed-sequence study is designed to evaluate the effect of multiple-dose Itraconazole or Rifampicin Capsules on the single-dose PK profiles of IMP4297 Capsules in healthy Chinese subjects.

32 subjects are planned to be enrolled (at least 12 subjects complete the study on one side).

Two parallel groups will be planned in this study with 16 subjects enrolled in each group. Two cycles are set for each group. The first group will be given IMP4297 and Itraconazole in a fixed sequence (two dosing regimens); The second group will receive IMP4297 and Rifampicin in a fixed sequence (two dosing regimens).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand the purpose, nature, methods and possible adverse reactions of the trial, voluntarily participate in the trial, and sign an informed consent form before any trial procedure, and promise to participate in all procedure of the trial.
2. Healthy Chinese male subjects aged 18 to 55 (inclusive) at the time of signing informed consent form.
3. Body mass index (BMI) ranges from 19.0 to 26.0 kg/m2 (inclusive); body weight ≥ 50.0 kg.
4. Subjects can communicate well with the investigators and understand and abide by the requirements of this trial.

Exclusion Criteria:

1. Subjects with past and present diseases with clinical abnormality in the opinion of the investigator, including but not limited to disease concerning nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolic system and skeletal system;
2. Subjects with allergic history (including drug and food allergies, etc.).
3. Subjects with history of dysphagia or any gastrointestinal disease that affects drug absorption judged by the investigator.
4. Subjects who have received surgery within 3 months before screening, or plan to have surgery during the trial period, or those who had surgery that will affects drug absorption (e.g. gastrectomy).
5. Subjects who cannot tolerate venipuncture, or have a history of needlesickness and fainting at the sight of blood.
6. Subject with lactose intolerability (who having had milk diarrhea).
7. Subjects who have drug abuse history within 6 months before screening, or have a positive urine drug screening (screening or baseline period) result.
8. Subjects who have used narcotics within 3 months before screening.
9. Subjects who consumed an average of more than 14 units of alcohol per week (1 unit of alcohol = 360 mL beer, 150 mL wine, or 45 mL liquor) within 3 months before screening, or who had a positive result of alcohol breath test (screening or baseline period), or could not give up alcohol during the trial.
10. Subjects who consumed an average of more than 5 cigarettes per day within 3 months before screening, or who could not stop using any tobacco products during the trial.
11. Subjects who consumed an average of excessive amounts of tea, coffee and / or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) every day within 3 months before screening.
12. Subjects who have participated in clinical trials of other study drugs/devices within 3 months before the first dose of the investigational drug, or have participated in 3 or more clinical trials of drugs/devices in the past year; if other study drugs have a longer half-life, the time interval will be longer and is required to be 5 half-lives of the drug.
13. Subjects who donated blood including blood component or have massive blood loss (2,200 mL), or received blood transfusion or used blood products within 3 months before screening.
14. Subjects who received vaccination within 4 weeks before screening.
15. Subjects who have taken any drugs [such as: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; SSRI antidepressants, cimetidine, macrolides, nitroimidazoles, sedative hypnotics, fluoroquinolones, antihistamines, antivirals (such as saquinavir), calcium antagonists (such as diltiazem, verapamil), rifamycins (such as rifampin)] that inhibit or induce the liver to metabolize drug within 28 days before the first dose of the investigational drug. If the past drug used has a longer half-life, the time interval will be longer and is required to be 5 half-lives of the drug, eg, Phenobarbital requires a 5-week washout period.
16. Subjects who have taken prescription drugs, over-the-counter drugs, dietary supplements or Chinese herbal medicine within 14 days before the first dose of the investigational drug. If the past drug used has a longer half-life, the time interval will be longer and is required to be 5 half-lives of the drug.
17. Any test result of hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody is positive.
18. At screening, vital signs (blood pressure, pulse and body temperature) examination, comprehensive physical examination and laboratory tests (hematology, blood biochemistry, urinalysis) indicate abnormal results with clinical significance according to the investigator. The reference normal range of vital signs (including the cut-off value) is as follows: Sitting systolic blood pressure is 90 to 139 mmHg, diastolic blood pressure is 60 to 89 mmHg, pulse is 50 to 100 bmp, body temperature (frontal temperature) is 36.0 to 37.0°C. The specific situation is comprehensively determined by the investigator.
19. At screening after a quiet rest for at least 10 min, the corrected QT interval (corrected by Fridericia's formula, QTcF = QT/RR1/3) > 450 msec or QRS complex > 120 msec was obtained by 12-lead ECG in supine position. If QTcF is more than 450 msec or QRS is more than 120 msec, 12-lead ECG measurement should be repeated twice, and the average value of QTcF or QRS measured three times is judged by the investigator as abnormality with clinical significance.
20. Subjects who are allergic to IMP4297, Itraconazole, Rifampicin, or to any ingredients of these preparations.
21. Vigorous exercise cannot be avoided within 48 hours before the first dose of the investigational drug and during the trial.
22. Subjects who consumed any food or beverages containing alcohol, caffeine, chocolate, or rich in xanthine within 48 hours before the first dose of the investigational drug; or those who cannot abstain from these products during the trial.
23. Subjects who cannot abstain from grapefruit or grapefruit-related citrus (eg, pomelo) or juice within 7 days before the first dose of investigational drug and during the trial;
24. Subjects or its partners who have birth plan, or are unwilling to adopt effective contraception methods (Annex 2), or have sperm donation plan throughout the trial and within 180 days after the last dose of the investigational drug.
25. Subjects who are unwilling or unable to follow the lifestyle guidelines described in the study protocol (such as dietary restrictions and activity requirements).
26. Subjects who have other acute or chronic medical or psychiatric diseases, which may increase the risks of participating in this trial, or may interfere with the interpretation of the trial results, will be judged unsuitable to participate in this trial by the investigator.
27. Subjects judged by the investigator to be unsuitable for participation in the trial.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum concentration) | 3 months
  peak concentration
AUC0-last (Area under the curve from time 0 to the last time with quantifiable concentration) | 3 months
  AUC0-last area under the curve from time zero to the time with the last quantifiable concentration
AUC0-inf (Area under the curve from time 0 to infinity) | 3 months
  area under the curve from time zero to infinity

SECONDARY OUTCOMES:
Number of Participants with Adverse Events That Are Related to Treatment | 3 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03
Tmax (Time to reach maximum concentration) | 3 months
  time to reach Cmax
t½ (Elimination half-life) | 3 months
  elimination half-life
CL/F (Apparent clearance) | 3 months
  apparent clearance
Vz/F (apparent volume of distribution ) | 3 months
  apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Pingsheng Xu, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Impact Therapeutics, Inc., Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hu X, Hsieh CY, Zhang Y, Liu W, Xu S, Cai SX, Liu L, Zhang M, Shi H, Zhang H, Liu P, Li X, Xu P. Effect of a strong CYP3A4 inhibitor and inducer on the pharmacokinetics of senaparib (IMP4297) in healthy volunteers: A drug-drug interaction study. Br J Clin Pharmacol. 2023 Jun;89(6):1767-1779. doi: 10.1111/bcp.15624. Epub 2023 Jan 3. PMID 36458825